CLINICAL TRIAL: NCT07149220
Title: Safety and Chemopreventive Efficacy of Fenretinide Mucoadhesive System in Subjects With Premalignant Oral Intraepithelial Neoplasia (OIN) Lesions: In Conjunction With Pharmacokinetic Assessment in Healthy Subjects.
Brief Title: Fenretinide Mucoadhesive Patch: Evaluation of Oral Cancer Prevention Efficacy in Adults With Premalignant Oral Lesions.
Acronym: FMS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan R. Mallery, DDS, PhD, Professor and Chair, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SMFMS-001.2025; R01CA227273 (NIH)
Record Dates: First submitted 2025-08-18; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Oral Leukoplakia; Oral Dysplasia
Keywords: oral cancer prevention
MeSH Terms: conditions — Leukoplakia, Oral

STUDY DESIGN:
Intervention Model Description: All participants with premalignant oral epithelial lesions will receive the active, fenretinide-releasing mucoadhesive system. There is no placebo control for this early Phase Ib study.
Masking Description: The research scientist who will be conducting the LOH analyses will be blinded as to whether the sample is pre or post treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMS impact on premalignant oral epithelial lesions (Experimental): Evaluation of the impact of the fenretinide-releasing system on premalignant oral epithelial lesions
  Interventions: Drug: Mucoadhesive fenretinide-releasing system (FMS)

INTERVENTIONS:
Drug: Mucoadhesive fenretinide-releasing system (FMS) — All persons with premalignant oral epithelial lesions will receive active intervention. The intervention consists of b.i.d. application of the FMS to the premalignant lesion for a total of six weeks. Please note that the intervention title Drug and intervention titled Other are the same entity.

SUMMARY:
The goal of this clinical trial is to determine the effect of a mucoadhesive system that releases the vitamin A derivative, fenretinide (FMS), on precancerous surface epithelial (lining tissue inside your mouth) changes. Specifically, does application of the FMS induce specific changes: 1) reduction in the clinical size, 2) reduction in the histologic grade of precancerous changes (determined by microscopic examination), 3) reduce the nuclear LOH events (changes in copy number of key genes to prevent oral cancer).

The first part of this study entails a single FMS application to persons having their wisdom teeth removed. This study is done to confirm how long the FMS needs to remain in place to release the cancer-preventive agent.

Participants will: 1) Have the FMS applied over the impacted wisdom tooth for 15 minutes, 2) FMS is removed, saliva is collected, and blood is drawn from a vein in the arm. 3) Tissue overlying the impacted wisdom tooth is removed and analyzed.

The second, multi-FMS application entails patients who have precancerous oral surface epithelial changes. These patients will have: 1) a piece of the precancerous tissue removed (biopsy) and examined under a microscope to ensure the diagnosis. Blood is drawn from a vein in the arm., 2) One week after the biopsy, return to discuss the results. If the changes are precancerous, this person will be given FMS to apply to the site twice a day. 3) Patients return every 7 to 10 days (for a total of six weeks) for an oral exam and clinical pictures, return the FMS, and obtain new FMS for the upcoming week., 4) At week 3 (midway), blood is drawn from a vein in the arm., 5) After the six weeks of treatment, clinical pictures are obtained, blood is drawn from a vein in the arm and all of the remaining treated tissue is completely removed. The patient is securely contacted and results are discussed. 6) Approximately 6 weeks after the final surgery, patients return for a complete oral examination and clinical pictures are obtained.

DETAILED DESCRIPTION:
1 Protocol Summary Overall Design The initial single patch application pharmacokinetic analysis on persons undergoing elective oral surgical procedures (third molar extraction) is being conducted to determine the requisite length of patch application time needed to achieve the predetermined fenretinide levels (0.1-3.0 µM) at the target tissue oral epithelium site.

Potential participants will be recruited during their mandatory pretreatment screening examination. Persons interested in participation will undergo informed consent. A single fenretinide patch will be applied to the oral mucosa overlying an impacted mandibular third molar and left in place for 15 minutes. Saliva and sera samples will be obtained immediately following patch removal. The treated oral mucosa will then be removed as the initial part of their surgical procedure for removal of a bony impacted third molar. If a 15-minute application is not sufficient to deliver the target fenretinide level in all 5 participants, subsequent participants (n=3) will be consented for a modified patch application time.

The multi-dose, investigator-initiated, single center, active formulation-only investigation is designed to assess the chemopreventive efficacy of a mucoadhesive fenretinide patch on microscopically confirmed premalignant oral epithelial lesions (oral intraepithelial neoplasia, OIN). Prospective patients will be recruited from persons with clinical lesions suspicious for OIN that are referred to Ohio State's College of Dentistry for management. We also have a large patient cohort (>200) of persons who are on long term follow up due to a previous diagnosis of premalignant oral epithelial lesions. Following the consultation and informed consent appointment, all participants will have an initial incisional biopsy of the lesion and this tissue will be used to establish baseline pretreatment parameters (histopathologic diagnosis and loss of heterozygosity indices). A diagnosis of premalignant oral epithelial disease (mild, moderate or severe epithelial dysplasia) is necessary to enter the chemoprevention study. Any person with advanced disease (i.e., oral squamous cell carcinoma) will be referred immediately for definitive care.

As this study will evaluate a novel drug delivery system, patients will be closely monitored (every 7 to 10 days) throughout the six-week fenretinide patch treatment period. At every recall appointment, a complete intraoral examination will be conducted and clinical images of the OIN lesion obtained. Participants will be instructed to return their used patches and additional fenretinide patches will be dispensed for the current treatment period. Random appointment saliva samples (2 over the treatment course) will be obtained for cotinine analyses to confirm no tobacco use. Sera samples will be obtained at the initial biopsy appointment and the final active study appointment (when the remaining OIN lesional tissue is excised). Patients will be given an after-hours call number and if complications arise, they will be instructed to discontinue patch administration and come to the clinical trial site for an evaluation the next day.

Following the six-week treatment course, the remaining OIN lesional tissue will be excised. Participants will be reappointed one week following the excisional biopsy to monitor healing and to discuss the final histopathologic biopsy results. All participants will be seen at a final recall appointment (approximately 6 weeks after cessation of treatment) during which time an intraoral examination and clinical image of treated OIN lesional site will be obtained. Instructions regarding the need to obtain follow up care will be provided.

1.1 Synopsis Title: Safety and Chemopreventive Efficacy of Fenretinide Mucoadhesive System in Subjects with Premalignant Oral Intraepithelial Neoplasia (OIN) Lesions; Preceded by Single Dose Pharmacokinetic Assessment in Healthy Subjects to Determine Application Time.

Study Description: A single 6.25 cm2 (12 mg fenretinide) mucoadhesive system (MS) pharmacokinetic analyses of target tissue (surface oral epithelium) from healthy subjects undergoing impacted mandibular third molar extraction to determine fenretinide patch application time necessary to achieve desired single dose drug level (0.1 to 3.0 µM fenretinide). Saliva and sera will also be obtained to assess drug absorption characteristics. 15-minute application time will be evaluated first; if tissue levels are insufficient, 30-minute application time will be evaluated. If 15-minute tissue levels exceed target, reduced application time will be pursued.

When application time is defined, a multi-dose clinical evaluation will proceed to determine chemopreventive efficacy of the fenretinide mucoadhesive system (FMS) on microscopically confirmed premalignant oral epithelial lesions (OIN, oral intraepithelial neoplasia).

Subjects will be trained in twice daily self-application of the FMS following mirror-guided patch placement. Subjects will be instructed to sit upright for the duration of their patch application.

Subjects will return to the study site every 7-10 days for 6 weeks to return used mucoadhesive systems and undergo applicable assessments.

Description of Study Intervention:

* Single Dose Pharmacokinetic Assessment in Healthy Subjects: Participants will be recruited at the mandatory screening appointment prior to their third molar surgery. A single 6.25 cm2 FMS (12 mg fenretinide) will be placed on the oral mucosa overlying the impacted mandibular third molar. Following a 15-minute application, the FMS will be removed, saliva and sera will be obtained, and the tissue underlying the patch excised to provide surgical access to the impacted third molar.
* Multi-dose Chemoprevention Evaluation in Subjects with OIN: Participants will apply the FMS to their OIN lesion, leave in place for 15 minutes, then remove and save the FMS to document use. This process will occur twice daily.

Study Duration:

* Single Dose Pharmacokinetic Assessment in Healthy Subjects: The anticipated study duration for accrual of five single-dose healthy subjects is approximately 2 months.
* Multi-dose Chemoprevention Evaluation in Subjects with OIN: The anticipated study duration for accrual of 25 multi-dose subjects with OIN is approximately 2 years, as funding permits.

Participant Duration:

* Single Dose Pharmacokinetic Assessment in Healthy Subjects: Individual participation is approximately 20 minutes.
* Multi-dose Chemoprevention Evaluation in Subjects with OIN: 6 weeks FMS application, 9 weeks/visits total Week/Visit 1: study explanation and consent; Week/Visit 2: incisional biopsy; Weeks/Visits 3-7: treatment (6 weeks, bid dosing, patient recall every 7 to 10 days); Week/Visit 8: recall appointment, excise remaining OIN tissue. Week/Visit 9: discuss final biopsy results, assess biopsy site healing. Visit 10, approximately six weeks post final biopsy. Clinical evaluation, provide instructions regarding need for follow up.

1.2 Schema

Single Dose Pharmacokinetic Assessment in Healthy Subjects:

1. All individuals undergoing elective third molar surgery must attend a consultation appointment. Potential study participants will be recruited during these consultation appointments. If the person is interested in study participation, the clinical trial will be discussed, and informed consent will be obtained.
2. Consented participants will arrive at their third molar surgical appointment 20 minutes prior to surgery to enable FMS placement and to obtain saliva and sera samples following FMS application. The overlying treated tissue will be removed as a portion of the third molar surgical procedure.

Multi-dose Chemoprevention Evaluation in Subjects with OIN:

1. Screen patient with suspicious oral lesion (white, white and red, or erythematous) tightly adherent, patch or plaque surface oral epithelial lesion with crisply delineated surface margins. Discuss clinical trial protocol, and if potential participant is interested, obtain informed consent. Subjects will be informed about the no-smoking policy. If patient is a current smoker, they will be requested to stop smoking and return in 6 weeks for incisional biopsy.
2. Conduct pretreatment incisional biopsy of suspicious oral lesion.
3. Participant recall, discuss initial biopsy results. If the suspicious lesion is microscopically confirmed to be premalignant, the participant will be enrolled in the study. Saliva sample obtained; cotinine levels checked at baseline then randomly throughout the study. Participants will be recalled every 7 to 10 days throughout the 6-week treatment period. Subjects will return used fenretinide mucoadhesive systems and obtain new FMS for the next treatment period.
4. Examination and excisional biopsy of residual OIN lesion after 6-week treatment.
5. Re-evaluation one week from excisional biopsy to discuss biopsy results and assess biopsy site.

Final study clinical assessment, approximately six weeks from excisional biopsy appointment to evaluate site and discuss final study results and need for clinical follow up.

ELIGIBILITY:
Inclusion Criteria:

* - Inclusion Criteria:

  * Adults, 18 years or older, with microscopically confirmed OIN. Only one clinically measurable OIN lesion (> 3x3 mm) and capable of full coverage by the FMS with a small zone of extension (2.1 x 2.1 cm smaller FMS, 2.8 x 2.8 larger FMS) will be evaluated in this study. If multiple suspicious lesions are noted, the most clinically advanced lesion will be selected for treatment. The patient will be provided the option to have the other lesions biopsied (self-pay and/or insurance) at another appointment or to schedule with another provider for management.
  * No use of tobacco products 6 weeks prior to and during the 6-week study. (confirmed via random cotinine saliva tests for former tobacco users).
  * Available for follow-up evaluations (every 7-10 days during trial), amenable to full 6-week study participation, and 6-week post-study recall.
  * All men and reproductive aged women of child bearing potential must agree to use contraception during treatment and 1 month after end of treatment. All reproductive aged, heterosexually active women must undergo monthly pregnancy testing.
  * Capable of providing informed consent.

Exclusion Criteria:

* - Exclusion Criteria:

  * Previous history of OSCC.
  * Microscopic diagnosis of OSCC or carcinoma in situ at the pretreatment biopsy.
  * Undergoing cancer treatments except for basal cell carcinoma of the skin.
  * Inability to stop tobacco product use.
  * Incapable of providing informed consent.
  * Pregnancy or unwilling to comply with birth control and monthly pregnancy testing criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Histopathologic grade (assessed using light microscopy) | The time frame is 12 months for participant recruitment and completion of the six week clinical trial.
  Complementary outcome measures of the Multi-dose Chemoprevention Evaluation in Subjects with OIN described separately. To evaluate both intra-participant (pretreatment and post treatment parameters) and collective assessments (all pretreatment findings relative to all post treatment findings) of the following chemoprevention indicators: Pretreatment and posttreatment lesional histologic grade, which will be determined by a ABOMP certified pathologist using light microscopy.
Clinical size (determined by measurement with a flexible ruler) | The time frame is 12 months for participant recruitment and completion of the six week clinical trial.
  Clinical images including internal measurement device (flexible ruler) to be taken prior to biopsy, and weekly at every monitoring visit.
Loss of heterozygosity (measured by genomic analyses | The time frame is 12 months for participant recruitment and completion of the six week clinical trial.
  Loss of heterozygosity indices at tumor suppressor gene loci associated with progression of OIN lesions to OSCC [3p14 (FHIT), 9p21 (INK4a/ARF), 9p22 (IFN-α), and 17p13 (p53)] (FHIT, p53, p16)] will be evaluated in DNA isolated from lesional epithelium.

SECONDARY OUTCOMES:
CYP4A4 and UGT1A1 enzyme levels (measured by image analysis quantified immunohistochemistry) | The time frame is 12 months for participant recruitment and completion of the six week clinical trial.
  Immunohistochemical staining to evaluate levels of fenretinide relevant enzymes (CYP4A4 and UGT1A1) in pre and post treatment biopsy specimens, quantified by image analysis.
fenretinide patch acceptance (measured by validated assessment tool completed by patients) | The time frame is 12 months for participant recruitment and completion of the six week clinical trial.
  Use a validated assessment tool to determine patient acceptability with regard to fenretinide patch adherence and residual after taste.

CONTACTS AND LOCATIONS:
Overall Officials: Susan R. Mallery, DDS, PhD, Principal Investigator — Ohio State University College of Dentistry
Locations (1):
- Ohio State University College of Dentistry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
While individual participant responsiveness will be reported in our publications, these data will be coded and therefore not identifiable with regard to the particular individual. We do not intend to report an HIPAA associated data.

REFERENCES:
- [Background] Desai KG, Mallery SR, Holpuch AS, Schwendeman SP. Development and in vitro-in vivo evaluation of fenretinide-loaded oral mucoadhesive patches for site-specific chemoprevention of oral cancer. Pharm Res. 2011 Oct;28(10):2599-609. doi: 10.1007/s11095-011-0489-3. Epub 2011 Jun 15. PMID 21674264
- [Background] Wu X, Desai KG, Mallery SR, Holpuch AS, Phelps MP, Schwendeman SP. Mucoadhesive fenretinide patches for site-specific chemoprevention of oral cancer: enhancement of oral mucosal permeation of fenretinide by coincorporation of propylene glycol and menthol. Mol Pharm. 2012 Apr 2;9(4):937-45. doi: 10.1021/mp200655k. Epub 2012 Mar 6. PMID 22280430
- [Background] Holpuch AS, Phelps MP, Desai KG, Chen W, Koutras GM, Han BB, Warner BM, Pei P, Seghi GA, Tong M, Border MB, Fields HW, Stoner GD, Larsen PE, Liu Z, Schwendeman SP, Mallery SR. Evaluation of a mucoadhesive fenretinide patch for local intraoral delivery: a strategy to reintroduce fenretinide for oral cancer chemoprevention. Carcinogenesis. 2012 May;33(5):1098-105. doi: 10.1093/carcin/bgs122. Epub 2012 Mar 15. PMID 22427354
- [Background] Wang D, Pei P, Shea F, Spinney R, Chang A, Lahann J, Mallery SR. Growth modulatory effects of fenretinide encompass keratinocyte terminal differentiation: a favorable outcome for oral squamous cell carcinoma chemoprevention. Carcinogenesis. 2024 Jun 10;45(6):436-449. doi: 10.1093/carcin/bgae022. PMID 38470060
- See also: URL for Desai et al. publication — https://pubmed.ncbi.nlm.nih.gov/21674264/
- See also: URL for the Holpuch et al. publication — https://pubmed.ncbi.nlm.nih.gov/22427354/
- See also: URL for the Wu et al. publication — https://europepmc.org/article/MED/22280430